CLINICAL TRIAL: NCT01142570
Title: Effect of Enteral Nutrition Enriched in Protein and Based on Indirect Calorimetry Measurement in Chronically Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Beit Rivka Hospital (Unknown)
Responsible Party: Dr. Papirov Gregory, Beit Rivka Hospital , Geriatric medical center, Petah Tikva, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5668
Record Dates: First submitted 2010-05-13; First posted 2010-06-11 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-01

CONDITIONS: Critically Ill
Keywords: Mechanical Ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Active Comparator): Patients will be receive caloric support as dictated by Hariss-Benedict Formula (Group 1)
  Interventions: Other: Caloric Support (Group 1)
- Group 2 (Active Comparator): Patients will be receive caloric support as dictated by Indirect Calorimetry (Group 2)
  Interventions: Other: Caloric Support (Group 2)
- Group 1A (Active Comparator): After seven days of hospitalization and study enrollment patients who have not been weaned from ventilator, will be divided into three groups.
  Patients in the first(Group 1A)group will receive caloric support calculated by the HARISS BENEDICT equation and protein dose of 1.1 to 1.5 grams per kilogram weight.
  Interventions: Dietary Supplement: Protein dose of 1.1 to 1.5 grams per kilogram weight.
- Group 2A (Active Comparator): After seven days of hospitalization and study enrollment patients who have not been weaned from ventilator, will be divided into three groups.
  Patients in the second group(Group 2A) will receive caloric support as measured by indirect calorimetry and will receive protein at 1.1 grams per kilogram weight.
  Interventions: Dietary Supplement: Protein at 1.1 grams per kilogram weight.
- Group 3A (Active Comparator): After seven days of hospitalization and study enrollment patients who have not been weaned from ventilator, will be divided into three groups.
  Patients in the third group will receive caloric support as measured by indirect calorimetry and will receive protein at a dose of 1.5 grams per kilogram weight.
  Interventions: Dietary Supplement: protein at a dose of 1.5 grams per kilogram weight.

INTERVENTIONS:
Other: Caloric Support (Group 1) — Four group 1-dose of caloric support will be calculated by Hariss-Benedict Formula measurement of Resting Energy Expenditure(REE).
  Arms: Group 1
Other: Caloric Support (Group 2) — For group 2- dose of caloric support will be calculated by Indirect Calorimetric measurement of Resting Energy Expenditure(REE)
  Arms: Group 2
Dietary Supplement: Protein dose of 1.1 to 1.5 grams per kilogram weight. — Patients in the first group(Group 1A) will receive caloric support calculated by the HARRISS BENEDICT equation and protein dose of 1.1 to 1.5 grams per kilogram weight.
  Arms: Group 1A
Dietary Supplement: Protein at 1.1 grams per kilogram weight. — Patients in the second group(Group 2A) will receive caloric support as measured by indirect calorimetry and will receive protein at 1.1 grams per kilogram weight.
  Arms: Group 2A
Dietary Supplement: protein at a dose of 1.5 grams per kilogram weight. — Patients in the third group (Group 3A) will receive caloric support as measured by indirect calorimetry and will receive protein at a dose of 1.5 grams per kilogram weight.
  Arms: Group 3A

SUMMARY:
This is a single-center, prospective, randomized, comparative, double-blind controlled clinical study intended to establish 1) the optimal method of determining calorie requirements and 2) the optimal amount of protein supply in chronically ventilated patients.

DETAILED DESCRIPTION:
The study will be performed in a chronic ventilation department.

Enrolled patients will be randomly allocated to receive calories as dictated by:

The Harriss-Benedict formula (Group 1) or Indirect Calorimetry (Group 2)

After one week of admission to the hospital department and study enrollment we will review the first results of the study.

After seven days of hospitalization and study enrollment patients who have not been weaned from the ventilator, will be divided into three groups.

1. Patients in the first group will receive caloric support calculated by the HARRISS BENEDICT equation and protein dose of 1.1 to 1.5 grams per kilogram weight.
2. Patients in the second group will receive caloric support as measured by indirect calorimetry and will receive protein at 1.1 grams per kilogram weight.
3. Patients in the third group will receive caloric support as measured by indirect calorimetry and will receive protein at a dose of 1.5 grams per kilogram weight.

Outcome of treatment results will be performed after one ,four and eight weeks:

1. Length of hospitalization
2. Weaning from Mechanical Ventilation
3. Development and progression of pressure ulcers
4. Infectious diseases incidence
5. Amount of insulin needed for glucose control
6. Length of mechanical ventilation
7. Readmission to Intensive Care Unit
8. Mortality rate

ELIGIBILITY:
Inclusion Criteria:

* Chronically Mechanical Ventilated Patients (more than 21 days of Mechanical Ventilation) by tracheostomy,
* Between ages 65-90

Exclusion Criteria:

* Patient over age 90 and younger the age of 65
* PH level less than 7.3 due to metabolic causes.
* A patient with blood albumin level less than 2.2 g / dl

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Successful weaning from ventilation | At one, four and eight weeks
  Spontaneous breathing
Length of hospital stay | At 8 weeks
  Length of hospitalization, in days
Readmission to Intensive Care Unit | At four and eight weeks.
Readmission to Intensive Care Unit Mortality | At eight weeks
Length of mechanical ventilation | At one, four and eight weeks
  Length of mechanical ventilation in days/hours

SECONDARY OUTCOMES:
Infectious diseases incidence | At one, four and eight weeks
Development and progression of pressure ulcers | At one, four and eight weeks
Checked daily insulin intake among different groups of patients | After one, four and eight weeks
  Glucose Control

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Papirov, MD, Principal Investigator — Beit- Rivka Hospital, Petah-Tikva, Israel; Pierre Singer, MD, Professor, Study Director — ICU, Rabin Medical Center,Petah- Tikva, Israel; Ludmila Zaidenberg, MD, Study Director — Beit Rivka hospital, Petah- Tikva, Israel; Milana Grinev, RN,Study Coordinator, Study Director — ICU, Rabin Medical Center,Petah- Tikva, Israel